CLINICAL TRIAL: NCT00173628
Title: Autoantibodies in Patients With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700824
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood drawing

SUMMARY:
Evaluate the autoantibodies, such as glutamic acid decarboxylase (GAD65), tyrosine phosphatase (IA-2 or ICA125), islet autoantibodies (IAA) and other associated autoimmune autoantibodies: microsomal antibodies, thyroglobulin antibodies, gastric parietal cell antibodies in patients with type 1 DM.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (DM) is a common disease in pediatric endocrine clinic and epidemiological studies showed the racial variation in the incidence, with the highest of 35 cases per 100000 in Finland. The incidence of type 1 DM in Taiwan is reported to be 1.5 per 100000 for the population less than 30 years old. While the diagnosis is made, the residual islet cell function is only about 20% of normal population. Therefore, the principle therapy in these patients is insulin therapy lifelong.

The pathogenesis of type 1 diabetes mellitus is multifactorial and controversial, involving the genetic and environmental factors. Type 1 DM is an autoimmune disease, which is T cell mediated islet cell destruction. Ninety percent of patients with type 1 DM express at least one of the autoantibodies to the islet. Antibodies to glutamic acid decarboxylase 65 (GAD65) were observed in 60-80% of such patients, which were considered the most important autoantigens. The autoantibodies disappeared successively after diagnosis and decreased in concentrations over time, but titers of antibodies to GAD65 had been observed fluctuated in patients with type 1 DM.

The prevalence of GAD antibodies, insulin autoantibodies, IA-2 (tyrosine phosphatase) were reported as 45-67%, 23-67% and 49%, respectively in Taiwan. Other associated autoimmune disease, such as autoimmune thyroiditis were reported as 13-24%. Such differences may be caused by the enrolling criteria and different age population. Therefore, we want to elucidate the role of autoantibodies in the pathogenesis of type 1 DM.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with type 1 diabetes

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150
Dates: Start 1990-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ching Tung, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan